CLINICAL TRIAL: NCT00829829
Title: A Multi-Center, Randomized, Double-Blind, Placebo Controlled Study of the Efficacy and Safety of Rilonacept for the Prophylaxis of Gout Flares During the Initiation of Allopurinol Therapy
Brief Title: PREventative Study Against URate-lowering Drug-induced Gout Exacerbations 1
Acronym: PRE-SURGE1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IL1T-GA-0810
Record Dates: First submitted 2009-01-23; First posted 2009-01-27 (Estimated); Results first posted 2017-04-28 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-03

CONDITIONS: Intercritical Gout
Keywords: Metabolism, Inborn Errors; Allopurinol; Metabolic Diseases; Genetic Diseases, Inborn; Musculoskeletal Diseases; Joint Diseases; Arthritis; Rheumatic Diseases; Metabolic disorder; Purine-Pyrimidine Metabolism, Inborn Errors; Gout
MeSH Terms: conditions — Metabolism, Inborn Errors; Metabolic Diseases; Genetic Diseases, Inborn; Musculoskeletal Diseases; Joint Diseases; Arthritis; Rheumatic Diseases; Purine-Pyrimidine Metabolism, Inborn Errors; Gout | interventions — rilonacept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Placebo (Placebo Comparator): Two subcutaneous injections of Placebo (for Rilonacept) as a loading dose on Day 1 followed by a single injection once a week (qw) from Week 1 to Week 15.
  Interventions: Other: Placebo
- Rilonacept 80 mg (Active Comparator): Two subcutaneous injections of Rilonacept 80 mg (for a total of 160 mg) as a loading dose on Day 1, followed by a single 80 mg injection of Rilonacept qw from Week 1 to Week 15.
  Interventions: Drug: Rilonacept 80 mg
- Rilonacept 160 mg (Active Comparator): Two subcutaneous injections of Rilonacept 160 mg (for a total of 320 mg) as a loading dose on Day 1, followed by a single 160 mg injection of Rilonacept qw from Week 1 to Week 15.
  Interventions: Drug: Rilonacept 160 mg

INTERVENTIONS:
Other: Placebo — Placebo loading dose followed by placebo injections (2 mL) qw for 16 weeks.
  Arms: Placebo
Drug: Rilonacept 80 mg — Rilonacept 160 mg loading dose followed by Rilonacept 80 mg/2 mL injections qw for 16 weeks.
  Arms: Rilonacept 80 mg
Drug: Rilonacept 160 mg — Rilonacept 320 mg loading dose followed by Rilonacept 160 mg/2 mL injections qw for 16 weeks.
  Arms: Rilonacept 160 mg

SUMMARY:
The purpose of this clinical research study was to determine the safety and effectiveness of an experimental drug called rilonacept in subjects with gout who are beginning allopurinol treatment for gout. Subjects will participate in this study for approximately 22 weeks. Rilonacept is being studied for use in preventing allopurinol-induced gout flares.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 to 80 years of age;
* Previously met the preliminary criteria of the American Rheumatism Association (ARA) for the classification; of the acute arthritis of primary gout;
* At least 2 gout flares in the year prior to the screening visit;
* Serum uric acid greater than or equal to 7.5 mg/dL at the screening visit;

Exclusion Criteria:

* Acute gout flare within 2 weeks of the screening visit or during screening;
* Persistent chronic or active infections;
* History of an allergic reaction to allopurinol;
* History or presence of cancer within 5 years of the screening visit;
* Previous exposure to Rilonacept;
* Use of allopurinol, benzbromarone, febuxostat, probenecid or sulfinpyrazone within 3 months prior to the screening visit.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2009-02; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (87):
- United States (64):
  - Birmingham, Alabama
  - Gilbert, Arizona
  - Peoria, Arizona
  - Searcy, Arkansas
  - Concord, California
  - San Diego, California
  - Santa Maria, California
  - Trumball, Connecticut
  - Washington D.C., District of Columbia
  - Daytona Beach, Florida
  - Delray Beach, Florida
  - Jacksonville, Florida
  - Jupiter, Florida
  - Naples, Florida
  - St. Petersburg, Florida
  - Gainsville, Georgia
  - Rome, Georgia
  - Tucker, Georgia
  - Woodstock, Georgia
  - Boise, Idaho
  - Avon, Indiana
  - Evansville, Indiana
  - South Bend, Indiana
  - Wichita, Kansas
  - Bowling Green, Kentucky
  - Owensboro, Kentucky
  - Baltimore, Maryland
  - Ellicott City, Maryland
  - Resistertown, Maryland
  - Troy, Michigan
  - Jackson, Mississippi
  - Florissant, Missouri
  - Las Vegas, Nevada
  - Berkeley Heights, New Jersey
  - Freehold, New Jersey
  - Brooklyn, New York
  - Greensboro, North Carolina
  - Hickory, North Carolina
  - Morehead City, North Carolina
  - Raleigh, North Carolina
  - Salisbury, North Carolina
  - Akron, Ohio
  - Cincinnati, Ohio
  - Middleburg Heights, Ohio
  - Perrysburg, Ohio
  - Duncansville, Pennsylvania
  - Fountain Hill, Pennsylvania
  - Huntingdon Valley, Pennsylvania
  - Lancaster, Pennsylvania
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Greer, South Carolina
  - North Charleston, South Carolina
  - Rock Hill, South Carolina
  - Memphis, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - Longview, Texas
  - Richardson, Texas
  - San Antonio, Texas
  - Burke, Virginia
  - Richmond, Virginia
  - Spokane, Washington
  - Tacoma, Washington
- Canada (23):
  - Calgary, Alberta
  - Burnaby, British Columbia
  - Kamloops, British Columbia
  - Kelowna, British Columbia
  - Quesnel, British Columbia
  - Victoria, British Columbia
  - Mount Pearl, Newfoundland and Labrador
  - St. John's, Newfoundland and Labrador
  - Brampton, Ontario
  - Corunna, Ontario
  - Fort Erie, Ontario
  - Greater Sudbury, Ontario
  - Kitchener, Ontario
  - Listowel, Ontario
  - London, Ontario
  - Mississauga, Ontario
  - Newmarket, Ontario
  - Toronto, Ontario
  - Windsor, Ontario
  - Montreal, Quebec
  - Québec, Quebec
  - Trois-Rivières, Quebec
  - Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Schumacher HR Jr, Evans RR, Saag KG, Clower J, Jennings W, Weinstein SP, Yancopoulos GD, Wang J, Terkeltaub R. Rilonacept (interleukin-1 trap) for prevention of gout flares during initiation of uric acid-lowering therapy: results from a phase III randomized, double-blind, placebo-controlled, confirmatory efficacy study. Arthritis Care Res (Hoboken). 2012 Oct;64(10):1462-70. doi: 10.1002/acr.21690. PMID 22549879
- See also: Rilonacept — http://druginfo.nlm.nih.gov/drugportal/ProxyServlet?mergeData=true&objectHandle=DBMaint&APPLICATION_NAME=drugportal&actionHandle=default&nextPage=jsp/drugportal/ResultScreen.jsp&TXTSUPERLISTID=501081761&QV1=RILONACEPT
- See also: Allopurinol — http://druginfo.nlm.nih.gov/drugportal/ProxyServlet?mergeData=true&objectHandle=DBMaint&APPLICATION_NAME=drugportal&actionHandle=default&nextPage=jsp/drugportal/ResultScreen.jsp&TXTSUPERLISTID=000315300&QV1=ALLOPURINOL
- See also: Allopurinol sodium — http://druginfo.nlm.nih.gov/drugportal/ProxyServlet?mergeData=true&objectHandle=DBMaint&APPLICATION_NAME=drugportal&actionHandle=default&nextPage=jsp/drugportal/ResultScreen.jsp&TXTSUPERLISTID=017795210&QV1=ALLOPURINOL+SODIUM

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 49 study sites in Unites States (US) and 15 study sites in Canada between 5 March 2009 and 18 May 2010. A total of 468 participants were screened in the study.
Pre-assignment Details: Out of 468 participants, 241 were randomized and 240 treated in the study. Participants were randomized in 1:1:1 ratio to receive either Placebo or Rilonacept 80 mg or Rilonacept 160 mg.
Groups:
- Placebo: Two subcutaneous injections of Placebo (for Rilonacept ) as a loading dose on Day 1 followed by a single injection once a week (qw) from Week 1 to Week 15.
Period: Overall Study
Arm/Group | Placebo | Rilonacept 80 mg | Rilonacept 160 mg
Started | 80 | 80 | 81
Treated (Participants treated were included in safety population.) | 79 | 80 | 81
Completed | 58 | 64 | 70
Not Completed | 22 | 16 | 11
Not completed — Protocol Violation | 0 | 3 | 0
Not completed — Adverse Event | 4 | 4 | 3
Not completed — Withdrawal by Subject | 8 | 4 | 2
Not completed — Decision by the Sponsor | 1 | 0 | 2
Not completed — Lost to Follow-up | 7 | 3 | 3
Not completed — Other than specified above | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Baseline population included full analysis set (FAS) comprising of all randomized participants who received any study medication and was based on treatment allocated by Interactive voice response system (IVRS) at randomization (as randomized).
Groups:
- Placebo: Two subcutaneous injections of Placebo (for Rilonacept ) as a loading dose on Day 1 followed by a single injection qw from Week 1 to Week 15.
- Total: Total of all reporting groups
Arm/Group | Placebo | Rilonacept 80 mg | Rilonacept 160 mg | Total
Number analyzed (Participants) | 79 | 80 | 81 | 240
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (13.6) | 52.9 (12.5) | 51.9 (11.6) | 52.3 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 9 | 5 | 17
  Male | 76 | 71 | 76 | 223
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 2 | 6
  Not Hispanic or Latino | 77 | 78 | 79 | 234
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 4 | 5 | 1 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 11 | 15 | 10 | 36
  White | 64 | 60 | 69 | 193
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Gout Flares Per Participant Assessed From Day 1 to Day 112 (Week 16)
Description: A gout flare was defined as participant reported acute articular pain typical of a gout attack that required treatment with an anti-inflammatory therapeutic: had at least 3 of the following 4 signs or symptoms: joint swelling, tenderness, redness, and pain and with at least 1 of the following: rapid onset of pain, decreased range of motion, joint warmth or other symptoms similar to a prior gout flare. Number of gout flares per participant was reported for this outcome measure. For drop-outs, only flares occurred before Day 112 were counted, regardless whether the flares occurred during the treatment period or not.
Time Frame: Day 1 to Day 112 (Week 16)
Population: Full analysis set (FAS) that included all randomized participants who received any study medication and was based on the treatment allocated by IIVRS at randomization (as randomized).
Measure: Mean (Standard Deviation); unit: Number of Gout flares per participant
Arm/Group | Placebo | Rilonacept 80 mg | Rilonacept 160 mg
Number analyzed (Participants) | 79 | 80 | 80
Number of Gout flares per participant | 1.06 (1.59) | 0.29 (0.77) | 0.21 (0.54)

2. Secondary Outcome: Number of Modified Gout Flares Per Participant From Day 1 to Day 112 (Week 16)
Description: Modified gout flare was defined using modified definition of a gout flare as participant-reported articular pain typical of a gout attack that was deemed to require treatment with anti-inflammatory therapy. Number of modified gout flares per participant were reported for this outcome measure.
Time Frame: Day 1 to Day 112 (Week 16)
Population: Full analysis set (FAS) that included all randomized participants who received any study medication and was based on the treatment allocated by IVRS at randomization (as randomized).
Measure: Mean (Standard Deviation); unit: modified gout flares
Arm/Group | Placebo | Rilonacept 80 mg | Rilonacept 160 mg
Number analyzed (Participants) | 79 | 80 | 80
modified gout flares | 1.19 (1.75) | 0.40 (0.91) | 0.28 (0.62)

3. Secondary Outcome: Percentage of Participants With at Least One Gout Flare From Day 1 to Day 112 (Week 16)
Description: Gout flare was defined as acute articular pain typical of a gout attack that required treatment with an anti-inflammatory therapeutic: had at least 3 of the following 4 signs or symptoms: joint swelling, tenderness, redness, and pain; and with at least 1 of the following: rapid onset of pain, decreased range of motion, joint warmth or other symptoms similar to a prior gout flare. Percentage of participants with at least one gout flare was reported for this outcome measure.
Time Frame: Day 1 to Day 112 (Week 16)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Rilonacept 80 mg | Rilonacept 160 mg
Number analyzed (Participants) | 79 | 80 | 81
percentage of participants | 46.8 | 18.8 | 16.3

4. Secondary Outcome: Percentage of Participants With at Least Two Gout Flares From Day 1 to Day 112 (Week 16)
Description: Gout flare was defined as acute articular pain typical of a gout attack that required treatment with an anti-inflammatory therapeutic: had at least 3 of the following 4 signs or symptoms: joint swelling, tenderness, redness, and pain, and with at least 1 of the following: rapid onset of pain, decreased range of motion, joint warmth or other symptoms similar to a prior gout flare. Percentage of participants with at least two gout flares was reported for this outcome measure.
Time Frame: Day 1 to Day 112 (Week 16)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Rilonacept 80 mg | Rilonacept 160 mg
Number analyzed (Participants) | 79 | 80 | 81
percentage of participants | 31.6 | 5.0 | 3.8

5. Secondary Outcome: Number of Gout Flare Days Per Participant From Day 1 to Day 112 (Week 16)
Description: Gout flare was defined as acute articular pain typical of a gout attack that required treatment with an anti-inflammatory therapeutic: had at least 3 of the following 4 signs or symptoms: joint swelling, tenderness, redness, and pain, and with at least 1 of the following: rapid onset of pain, decreased range of motion, joint warmth or other symptoms similar to a prior gout flare. Number of gout flare days per participant was reported for this outcome measure.
Time Frame: Day 1 to Day 112 (Week 16)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Gout flare Days
Arm/Group | Placebo | Rilonacept 80 mg | Rilonacept 160 mg
Number analyzed (Participants) | 79 | 80 | 80
Gout flare Days | 5.52 (9.73) | 2.36 (11.35) | 0.98 (2.95)

6. Secondary Outcome: Number of Gout Flare Days With Participant's Pain Score of 5 or More (From Daily Diary) Per Participant From Day 1 to Day 112 (Week 16)
Description: Participants were asked to complete a telephone diary by calling the IVRS daily beginning at the baseline visit (Day 1) through the follow-up visit (Day 141) and reported their general well-being, gout symptoms, and weekly study drug administrations. At the onset of pain from a gout flare, participants were to answer additional diary questions regarding their gout flare and had to continue daily flare assessments until they reported the flare had ended. If a flare occurred just prior to the follow-up visit (Day 141), participants were to continue completing the daily diary until the flare resolved. Gout flare pain was assessed on a scale from 0 to 10 (with 0=no pain and 10=severe pain) within the past 24 hours.
Time Frame: Day 1 to Day 112 (Week 16)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Gout flare days
Arm/Group | Placebo | Rilonacept 80 mg | Rilonacept 160 mg
Number analyzed (Participants) | 79 | 80 | 80
Gout flare days | 2.13 (3.20) | 0.85 (3.93) | 0.35 (1.30)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from signature of the informed consent form up to the final visit (Week 20) regardless of seriousness or relationship to investigational product.
Description: Reported adverse events are treatment-emergent adverse events that is AEs that developed/worsened during the 'on treatment period' (time from the administration of first dose of study drug up to 35 days after the last dose of study drug). Analysis was performed on safety population included all participants who received any study medication and was based on the treatment received.
Arm/Group | Placebo | Rilonacept 80 mg | Rilonacept 160 mg
Serious Adverse Events (participants affected / at risk) | 3/79 | 3/80 | 3/81
Other Adverse Events (participants affected / at risk) | 8/79 | 16/80 | 17/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=79) | Rilonacept 80 mg (N=80) | Rilonacept 160 mg (N=81)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal hernia obstructive (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=79) | Rilonacept 80 mg (N=80) | Rilonacept 160 mg (N=81)
Injection site erythema (General disorders) | 0 (0) | 4 (4) | 3 (9)
Injection site reaction (General disorders) | 0 (0) | 1 (1) | 5 (10)
Bronchitis (Infections and infestations) | 1 (1) | 4 (4) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 4 (4) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (6) | 2 (3) | 3 (3)
Headache (Nervous system disorders) | 1 (1) | 5 (6) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI/Institution will provide a copy of any publication to Sponsor prior to submission for review. Sponsor may request to remove confidential information from submission, provided that removal does not preclude the complete and accurate presentation and interpretation of the study results.